CLINICAL TRIAL: NCT00022646
Title: A Phase II Clinical Trial Evaluating Three Schedules Of ALIMTA Plus Gemcitabine As Frontline Chemotherapy For Patients With Locally Advanced Or Metastatic Non-Small Cell Lung Cancer
Brief Title: Pemetrexed Disodium Plus Gemcitabine in Treating Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0026; NCI-2012-02399 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000068838 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-08-10; First posted 2003-01-27 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I: pemetrexed + gemcitabine (Experimental): Patients receive pemetrexed disodium IV over 10 minutes on day 1 followed by gemcitabine IV over 30 minutes on days 1 and 8.
  Interventions: Drug: gemcitabine hydrochloride; Drug: pemetrexed disodium
- Arm II: pemetrexed + gemcitabine (Experimental): Patients receive gemcitabine IV over 30 minutes on days 1 and 8 followed by pemetrexed disodium IV over 10 minutes on day 1.
  Interventions: Drug: gemcitabine hydrochloride; Drug: pemetrexed disodium
- Arm III: pemetrexed + gemcitabine (Experimental): Patients receive gemcitabine IV over 30 minutes on day 1 and pemetrexed disodium IV over 10 minutes followed by gemcitabine IV over 30 minutes on day 8.
  Interventions: Drug: gemcitabine hydrochloride; Drug: pemetrexed disodium

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: pemetrexed disodium

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving more than one drug and giving the drugs in different ways may kill more tumor cells.

PURPOSE: Randomized phase II trial to compare the effectiveness of three different regimens of pemetrexed disodium plus gemcitabine in treating patients who have locally advanced or metastatic non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the tumor response rates in patients with locally advanced or metastatic non-small cell lung cancer treated with 3 different schedules of pemetrexed disodium and gemcitabine.
* Compare the duration of response, time to progressive disease, time to treatment failure, and survival time in patients treated with these regimens.
* Compare the quantitative and qualitative toxic effects of these regimens in these patients.

OUTLINE: This is a randomized, open-label study. Patients are stratified according to stage of disease (IIIB vs IV) and ECOG performance status (0 vs 1). Patients are randomized to one of three treatment arms.

* Arm I: Patients receive pemetrexed disodium IV over 10 minutes on day 1 followed by gemcitabine IV over 30 minutes on days 1 and 8.
* Arm II: Patients receive gemcitabine IV over 30 minutes on days 1 and 8 followed by pemetrexed disodium IV over 10 minutes on day 1.
* Arm III: Patients receive gemcitabine IV over 30 minutes on day 1 and pemetrexed disodium IV over 10 minutes followed by gemcitabine IV over 30 minutes on day 8.

Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease may receive up to 6 additional courses of therapy.

Patients are followed every 2 months for 1 year and then every 6 months for 4 years.

PROJECTED ACCRUAL: A total of 180 patients (60 per treatment arm) will be accrued for this study within 20 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed locally advanced or metastatic non-small cell lung cancer

  * Stage IIIB disease that is ineligible for combined modality therapy OR
  * Stage IV disease
* Measurable disease
* No clinically detectable (by physical exam) third-space fluid collection (e.g., ascites or pleural effusions) that cannot be controlled by drainage or other procedures
* No brain metastases (even if treated)

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9 g/dL

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST and ALT no greater than 3 times ULN (5 times ULN if liver metastases present)
* Alkaline phosphatase no greater than 3 times ULN (5 times ULN if liver metastases present)

Renal:

* Creatinine clearance at least 45 mL/min

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to take folic acid or cyanocobalamin (vitamin B12) supplementation
* No uncontrolled infection
* No concurrent chronic debilitating disease
* No weight loss of 10% or more within the past 6 weeks
* No other prior malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or noninvasive carcinoma

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior biologic or genetic therapy for lung cancer
* No concurrent immunomodulating agents

Chemotherapy:

* No prior chemotherapy for lung cancer

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy to a different site and recovered
* No prior radiotherapy to 25% or more of bone marrow
* No prior radiotherapy to whole pelvis
* No prior radiotherapy for primary disease
* No concurrent radiotherapy

Surgery:

* More than 4 weeks since prior major surgery

Other:

* No aspirin or nonsteroidal anti-inflammatory agents 2 days before, during, and for 2 days after pemetrexed disodium administration (5 days for long-acting agents such as piroxicam, naproxen, diflunisal, or nabumetone)
* No other concurrent cytostatic or cytotoxic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2001-08; Primary Completion 2003-11 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
tumor response rate | Up to 4 years

SECONDARY OUTCOMES:
duration of response | Up to 4 years
time to treatment failure | Up to 4 years
survival | Up to 4 years
time to disease progression | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Alex A. Adjei, MD, PhD, Study Chair — Mayo Clinic
Locations (22):
- United States (22):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Health Plaza, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota

REFERENCES:
- [Background] An MW, Mandrekar SJ, Branda ME, Hillman SL, Adjei AA, Pitot HC, Goldberg RM, Sargent DJ. Comparison of continuous versus categorical tumor measurement-based metrics to predict overall survival in cancer treatment trials. Clin Cancer Res. 2011 Oct 15;17(20):6592-9. doi: 10.1158/1078-0432.CCR-11-0822. Epub 2011 Aug 31. PMID 21880789
- [Background] Campbell ME, Mandrekar SJ, Hillman SL, et al.: What is the added value of actual tumor measurements (TM) in predicting overall survival (OS)? The North Central Cancer Treatment Group (NCCTG) findings. [Abstract] J Clin Oncol 26 (Suppl 15): A-6520, 2008.
- [Background] Jatoi A, Hillman S, Stella P, Green E, Adjei A, Nair S, Perez E, Amin B, Schild SE, Castillo R, Jett JR; North Central Cancer Treatment Group. Should elderly non-small-cell lung cancer patients be offered elderly-specific trials? Results of a pooled analysis from the North Central Cancer Treatment Group. J Clin Oncol. 2005 Dec 20;23(36):9113-9. doi: 10.1200/JCO.2005.03.7465. PMID 16361618
- [Result] Adjei AA, Salavaggione OE, Mandrekar SJ, Dy GK, Ziegler KL, Endo C, Molina JR, Schild SE, Adjei AA. Correlation between polymorphisms of the reduced folate carrier gene (SLC19A1) and survival after pemetrexed-based therapy in non-small cell lung cancer: a North Central Cancer Treatment Group-based exploratory study. J Thorac Oncol. 2010 Sep;5(9):1346-53. doi: 10.1097/JTO.0b013e3181ec18c4. PMID 20651609
- [Result] Ma CX, Nair S, Thomas S, Mandrekar SJ, Nikcevich DA, Rowland KM, Fitch TR, Windschitl HE, Hillman SL, Schild SE, Jett JR, Obasaju C, Adjei AA; North Central Cancer Treatment Group; Mayo Clinic; Eli Lilly & Company. Randomized phase II trial of three schedules of pemetrexed and gemcitabine as front-line therapy for advanced non-small-cell lung cancer. J Clin Oncol. 2005 Sep 1;23(25):5929-37. doi: 10.1200/JCO.2005.13.953. PMID 16135464